CLINICAL TRIAL: NCT03275610
Title: Risk Stratification Using Genetic Markers of Patients With a History of Pulmonary Embolism Post Total Hip or Total Knee Arthroplasty
Brief Title: Genetic Markers of Patients With History of Pulmonary Embolism Post Total Joint Arthroplasty
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Jay R. Lieberman, MD, Professor, University of Southern California
Other Study IDs: ORTHO-01
Record Dates: First submitted 2017-09-05; First posted 2017-09-07 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: Blood sample — 5 mL of blood withdrawn from patients with history of pulmonary embolism post total hip arthroplasty or total joint arthroplasty

SUMMARY:
This study seeks to uncover potential genetic determinants of pulmonary embolism (PE). Our translational goal is to ultimately identify certain genetic markers that will allow us to stratify patients in terms of their PE risk post total knee or total hip arthroplasty. The clinical implications for this study would allow for better patient care by lowering the risk of post-operative bleeding while still preventing symptomatic PEs and deep vein thromboses (DVTs). We look to sample patients who have a history of PE after undergoing total knee or total hip arthroplasty. We will sample these patients' blood DNA for a set of DNA genetic markers. To do so, we will utilize the Taqman assay, which is a PCR-based 5'-nuclease allelic discrimination assay to determine single nucleotide polymorphism (SNP) genotypes at specified loci. The region flanking the SNP is amplified using two allele-specific fluorescent probes, allowing for the detection of each allele in a single tube. Using this assay, there is no post-PCR processing because the probes are included in the PCR reaction (Hui). Using this approach, we will measure the frequency of genetic mutations in patients who have developed a PE after a total joint arthroplasty. This data would then be used to perform a prospective study to determine a subset of genetic markers that can definitively be used to risk stratify patients.

ELIGIBILITY:
Inclusion Criteria:

* patients with a history of Pulmonary Embolism and Total Hip Arthroplasty or Total Knee Arthroplasty, between the ages of 18 and 70 years

Exclusion Criteria:

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Established patients with a history of Pulmonary Embolism Post Total Hip Arthroplasty or Post Knee Arthroplasty
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-04-24 (Actual); Primary Completion 2026-04-23 (Estimated); Study Completion 2026-04-23 (Estimated)

PRIMARY OUTCOMES:
Identification of Genetic Mutations | 6 weeks Post Total Hip Arthroplasty or Post Total Knee Arthroplasty
  identify the frequency of genetic mutations in patients who have developed a PE after a total joint or total hip arthroplasty

CONTACTS AND LOCATIONS:
Overall Officials: Jay R Lieberman, MD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No